CLINICAL TRIAL: NCT02084277
Title: A Randomized Clinical Trial to Compare Oral Health Related Quality of Life Outcome for Patients With Malocclusion Receiving Orthodontic Treatment: Before Treatment vs. During Initial Treatment; Self-ligating Brackets vs. Conventional Brackets
Brief Title: A RCT to Compare OHRQoL Outcome for SLB and CB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Dr. Tai-ting Lai, Director of Orthodontic Department, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10MMHIS068
Record Dates: First submitted 2014-03-08; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Malocclusion
Keywords: Oral health-related quality of life (OHRQoL); Self-ligating brackets (SLB); Conventional brackets (CB); Oral Health Impact Profile-14 (OHIP-14); Short Form-36 (SF-36)
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-ligating brackets (Experimental): Several self-ligating brackets are currently FDA-approved but have not been rigorously studied in this malocclusion patient population or in comparison to traditional brackets methods. Unlike conventional brackets, Self-ligating brackets (SLB) are bracket systems, without the wire ligature or elastic ligature, that have a tube-like device build into the bracket to close off the edgewise slot.
  Interventions: Device: Self-ligating brackets (SLB)
- Conventional brackets (Placebo Comparator): The conventional brackets (CB) (edgewise appliance) retain the basic principle design of a rectangular wire in a rectangular slot. Archwire are tied to the bracket once placed in the slot with either elastometric ligation ties ("O-rings") or steel ligation.
  Interventions: Device: Conventional brackets (CB)

INTERVENTIONS:
Device: Self-ligating brackets (SLB)
  Other Names: Damon Q
  Arms: Self-ligating brackets
Device: Conventional brackets (CB)
  Other Names: OPAK
  Arms: Conventional brackets

SUMMARY:
The objective of this prospective study is to compare these two treatments (conventional brackets v.s. self-ligating brackets) in malocclusion to determine which treatment will provide the better oral health related quality of life (OHRQoL) outcomes for patients during the initial orthodontic treatment compared with pretreatment.

ELIGIBILITY:
Inclusion Criteria:

* malocclusion patients
* age between 12 to 40 years
* suitable for orthodontic treatment using either self-ligating brackets or conventional brackets.

Exclusion Criteria:

* Any surgery performed in the previous days,
* Previous temporomandibular joint arthrotomies,
* Fewer than 20 teeth total or fewer than 10 teeth in each arch,
* Unstable residence or travel restrictions,
* Periodontal disease judged to be severe by the surgeon,
* Pregnancy,
* Previous mandibular surgery, and
* Inability to follow instructions or the study protocol.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Patient Reported Outcome - Oral Health Related Quality of Life | one month

SECONDARY OUTCOMES:
Pain | one month

CONTACTS AND LOCATIONS:
Overall Officials: Tai-ting Lai, DrPH, Principal Investigator — Mackay Memorial Hospital,Taipei, Taiwan
Locations (1):
- Orthodontic Department of Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Allen PF, McMillan AS, Walshaw D, Locker D. A comparison of the validity of generic- and disease-specific measures in the assessment of oral health-related quality of life. Community Dent Oral Epidemiol. 1999 Oct;27(5):344-52. doi: 10.1111/j.1600-0528.1999.tb02031.x. PMID 10503795
- [Background] Bergius M, Kiliaridis S, Berggren U. Pain in orthodontics. A review and discussion of the literature. J Orofac Orthop. 2000;61(2):125-37. doi: 10.1007/BF01300354. English, German. PMID 10783564
- [Background] Cacciafesta V, Sfondrini MF, Ricciardi A, Scribante A, Klersy C, Auricchio F. Evaluation of friction of stainless steel and esthetic self-ligating brackets in various bracket-archwire combinations. Am J Orthod Dentofacial Orthop. 2003 Oct;124(4):395-402. doi: 10.1016/s0889-5406(03)00504-3. PMID 14560269
- [Background] Chen M, Wang DW, Wu LP. Fixed orthodontic appliance therapy and its impact on oral health-related quality of life in Chinese patients. Angle Orthod. 2010 Jan;80(1):49-53. doi: 10.2319/010509-9.1. PMID 19852639
- [Background] Choi WS, Lee S, McGrath C, Samman N. Change in quality of life after combined orthodontic-surgical treatment of dentofacial deformities. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Jan;109(1):46-51. doi: 10.1016/j.tripleo.2009.08.019. PMID 20123378
- [Background] Eberting JJ, Straja SR, Tuncay OC. Treatment time, outcome, and patient satisfaction comparisons of Damon and conventional brackets. Clin Orthod Res. 2001 Nov;4(4):228-34. doi: 10.1034/j.1600-0544.2001.40407.x. PMID 11683812
- [Background] Erdinc AM, Dincer B. Perception of pain during orthodontic treatment with fixed appliances. Eur J Orthod. 2004 Feb;26(1):79-85. doi: 10.1093/ejo/26.1.79. PMID 14994886